CLINICAL TRIAL: NCT06104891
Title: Radicle Recharge™: A Randomized, Double-blind, Placebo-controlled Trial Assessing the Immediate Effects of Non-caffeinated Supplements on Energy Levels and Associated Health Outcomes
Brief Title: Radicle Recharge: A Study of Health and Wellness Products on Energy Levels and Other Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-2317
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Energy; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth, then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Control 1 (Placebo Comparator): Recharge Product Form 1 - control
  Interventions: Dietary Supplement: Recharge Placebo Control 1
- Active Product 1 (Experimental): Recharge Product Form 2 - active product 1
  Interventions: Dietary Supplement: Recharge Active Study Product 1
- Active Product 2 (Experimental): Recharge Product Form 3 - active product 1
  Interventions: Dietary Supplement: Recharge Active Study Product 2
- Active Product 3 (Experimental): Recharge Product Form 4 - active product 1
  Interventions: Dietary Supplement: Recharge Active Study Product 3

INTERVENTIONS:
Dietary Supplement: Recharge Placebo Control 1 — Participants will use their Radicle Recharge Placebo Control 1 as directed for a period of 5 hours.
  Arms: Placebo Control 1
Dietary Supplement: Recharge Active Study Product 1 — Participants will use their Radicle Recharge Active Study Product 1 as directed for a period of 5 hours.
  Arms: Active Product 1
Dietary Supplement: Recharge Active Study Product 2 — Participants will use their Radicle Recharge Active Study Product 2 as directed for a period of 5 hours.
  Arms: Active Product 2
Dietary Supplement: Recharge Active Study Product 3 — Participants will use their Radicle Recharge Active Study Product 3 as directed for a period of 5 hours.
  Arms: Active Product 3

SUMMARY:
A randomized, double blind, placebo-controlled trial assessing the immediate impact of non-caffeinated supplements on energy levels and associated health outcomes

DETAILED DESCRIPTION:
This is a randomized, double blind. placebo-controlled study conducted with adult participants (study volunteers, citizen scientists), at least 21 years of age at the time of consent and attending the Supply Side West Meeting (SSW) this year.

Eligible participants will (1) endorse a desire for more energy and (2) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known contraindication or with well-established, significant safety concerns due to illness and/or medication(s) will be excluded. Participants that report a known allergy to any possible ingredient they may be exposed to in one of the study arms will be excluded.

Participants will take their assigned study product at a Radicle booth, after enrolling.

Participant reported outcomes (PROs) are collected electronically from eligible participants at baseline (before study product consumption, and for a period of 5 hours after consuming their study product.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, sexes, and gender identities
* Attending the Supply Side West meeting in person
* Able to read and understand English
* Endorses more energy as a primary desire
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Reports current enrollment in another clinical trial
* Reports a cardiac disease that presents an absolute contraindication and/or a significant safety concern with any of the study product ingredients.
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study products ingredients: Anticoagulants, chemotherapy, immunotherapy, medications that warn against grapefruit consumption, oral diabetic medications, or oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection
* Reports an allergy to any of the study products ingredients

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in energy | 5 hours
  Mean difference in energy score as assessed by Energy Visual Analog Scale (VAS) (scale 0 - 10; where 0 is no energy and 10 is more than enough energy)

SECONDARY OUTCOMES:
Change in cognitive function | 5 hours
  Mean difference in cognitive function score as assessed by Patient Reported Outcome Measurement System (PROMIS) Cognitive Function - Abilities 4A (scale 4-20; where lower scores correspond to worse cognitive function). Modified timing to, "since walking this morning"
Change in fatigue | 5 hours
  Mean difference in fatigue score as assessed by Fatigue VAS (scale 0 - 10; where 0 is no fatigue and 10 is completely exhausted)
Minimal clinically important difference (MCID) in energy | 5 hours
  Likelihood of experiencing MCID in energy score as assessed by Energy VAS
Minimal clinically important difference (MCID) in cognitive function | 5 hours
  Likelihood of experiencing MCID in cognitive function score as assessed by PROMIS Cognitive Function - Abilities 4A
Minimal clinically important difference (MCID) in fatigue | 5 hours
  Likelihood of experiencing MCID in fatigue score as assessed by Fatigue VAS

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com